CLINICAL TRIAL: NCT02853409
Title: Prospective Epidemiological Study to Determine the Variation in the Quality of Life of Patients With Locally Advanced and Metastatic Prostate Cancer (PROS-PROSQoLI Study)
Brief Title: Quality of Life of Patients With Locally Advanced and Metastatic Prostate Cancer
Acronym: PROS-PROSQoLI
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-92-52014-215
Record Dates: First submitted 2016-04-01; First posted 2016-08-02 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate possible changes in quality of life related to health (HRQL) in locally advanced and metastatic prostate cancer patients, after one year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥ 18 years old
* Symptomatic prostate cancer patients who present symptoms due to prostate cancer disease
* Capacity to comply with the protocol
* Patient with an expected survival > 12 months

Exclusion Criteria:

* Patients who are also participating in any other clinical study
* Patient with other malignant diseases, apart from prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Quality of life evolution, using the validated Prostate Cancer Specific Quality of Life Instrument (PROSQOLI) | 12 months

SECONDARY OUTCOMES:
Socio-demographic characteristics (percentage of patients (a) living married or living with a partner, (b) had completed primary studies, (c) retired or pensioners, (d) patients had a family history of PrCa) | 12 months
Anthropometric Characteristics - Body Mass Index | Baseline
Prostate-specific Antigen (PSA) | Baseline, 12 months
Testosterone level | Baseline, 12 months
Digital rectal examination | Baseline, 12 months
Percentage of patients who have undergone previous treatment (surgery, radiotherapy and hormonotherapy) | 12 months
Anxiety questionnaire (Hospital Anxiety and Depression scales-HAD) | 12 months
Change in general health status perception (from either patient or physician perspective) | 12 months
  Assessment of health in relation to Prostate Cancer, the options are: very good, quite good, slightly good, neither good nor bad, slightly bad, quite bad or very bad.
Quality of life using EQ-5D questionnaire | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (14):
- Spain (14):
  - Hospital Quirón Campo de Gibraltar, Cadiz
  - H. San Juan de Dios, Córdoba
  - Hospital Quiron Vizcaya, Erandio
  - H. Can Misses, Ibiza Town
  - Hospital San Juan de Dios, León
  - H. de Torrelodones, Madrid
  - H. Montepríncipe, Madrid
  - Hospital Quirón San Camilo, Madrid
  - Hospital San Rafael, Madrid
  - Hospital Quirón Marbella, Marbella
  - Hospital Parque San Antonio, Málaga
  - H. Infanta Sofía, San Sebastián de los Reyes
  - Hospital NISA, Seville
  - Hospital Sagrado Corazón, Seville